CLINICAL TRIAL: NCT05315973
Title: Personalized Fingertip Glucose Measurement With a Touch Sensor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We never were able to start this study, as an NDA agreement had been signed, after we had anticipated enrolling, preventing starting.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward Chao, Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 801468
Record Dates: First submitted 2022-03-15; First posted 2022-04-07 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensor group (Experimental)
  Interventions: Device: Testing sensor vs glucometer

INTERVENTIONS:
Device: Testing sensor vs glucometer — Will test accuracy of this sensor; there will be no intervention.

SUMMARY:
Self-testing of glucose by patients living with diabetes mellitus (DM) involves needles, which causes discomfort or inconvenience eventually lead to decreased willingness to perform such needle-based check-ups that are vital to DM management. While technology has evolved, currently there is no glucose monitoring device that is needle-free. The investigators are studying a glucose sensor that detects glucose non-invasively, from sweat on an individual's fingertip. As it has not yet been tested in individuals with DM, the team will examine its accuracy and acceptability in these patients. Results from this clinical trial could serve as the basis for further development of a non-invasive glucose sensor.

ELIGIBILITY:
Inclusion Criteria:

* An existing diagnosis of diabetes mellitus, either T1DM or T2DM, or any other type or etiology of diabetes
* Having a hemoglobin A1c < 9.0%, and taking medication for diabetes. Individuals will bring their own lab report.
* Ability to provide informed consent for participation.

Exclusion Criteria:

* Individuals without diabetes
* Uncontrolled medical conditions, including diabetes with a hemoglobin A1c > 9.0%, hypertension, heart, kidney, or liver failure.
* Those who cannot speak or read English. Participation will be limited to those who read and speak English, as this is a pilot study of a small number of participants, that will very unlikely offer the prospect of direct benefit from participating.
* Individuals who have frequent hypoglycemia, hypoglycemia unawareness, or who are at high risk for hypoglycemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Accuracy: glucose readings in mg/dL | 1 day
  Correlation of touch sensor glucose readings compared with glucometer measurements

SECONDARY OUTCOMES:
Acceptability: questionnaire ratings on a scale of 1-5, with 5 being the highest | 1 day
  ease of use, and any other comments to optimize the design and function of this sensor, as reported by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Chao, DO, Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: Yes
This will include all data collected in the study, sensor glucose readings, as well as glucometer measurements.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: approximately 10 yrs